CLINICAL TRIAL: NCT05259618
Title: Project ARRR, ALT Routinely Recorded Remotely: A Comparator Study of Liver Function Tests Using the Tasso+ to Venipuncture.
Brief Title: ALT Routinely Recorded Remotely: A Comparator Study of Liver Function Tests Using the Tasso+ to Venipuncture.
Acronym: ARRR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tasso Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TALT01-20
Record Dates: First submitted 2022-02-16; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Elevated Alanine Transaminase (ALT)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with elevated alanine transaminase (ALT): patients with alanine transaminase (ALT) > 3x upper limit of normal (ULN).
  Interventions: Other: Tasso+ SST

INTERVENTIONS:
Other: Tasso+ SST — alternative site blood sample collection.
  Other Names: Tasso+

SUMMARY:
A direct comparison study of blood samples collected using the Tasso+ device and venous blood samples in patients with elevated alanine transaminase (ALT).

DETAILED DESCRIPTION:
This is a prospective, non-blinded, multi-center study to be conducted within the USA. This study will consist of a single arm. Blood will be drawn from each subject, using two different collection methods: the Tasso+ device and the conventional venipuncture method. The results will be compared assess correlation between blood collected at home, by the patient, using the Tasso+ device and blood collected in the office using a Vacutainer (SST, Red Top tube) using venipuncture for alanine transaminase (ALT), aspartate aminotransferase (AST) and total bilirubin.

Participants can complete up to 3 visits and will include self-collected blood samples using the Tasso+ device at home on the day of visit 2 and visit 3.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be willing and able to provide written informed consent prior to study entry
2. Subject is ≥ 18 years of age.
3. Subject must meet the following criterion:

   known recent history of liver function abnormality and requiring follow-up Liver tests (including ALT>3XULN)
4. Subject must be willing and able to adhere to the assessments, study schedule, prohibitions and restrictions as described in the protocol.
5. Patients may be on any treatment / therapeutic clinical trial as indicated by treating physician

Exclusion Criteria:

1. Pregnant or nursing female by self-report.
2. Presents with abnormal skin integrity or atypical skin health within the areas to be tested (upper shoulders).
3. Subjects who have applied lotion to the skin on the shoulder the day of the visit.
4. Patients with hepatic encephalopathy
5. Vulnerable populations (children, prisoners, pregnant women, participants with diminished decision-making capacity, illiterate populations, educationally disadvantaged populations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an ALT > 3 X upper limit of normal
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Venous and Tasso+ blood sample comparison for ALT | through study completion, an average of 1 Year and 6 Months
  Correlation between blood collected at home, by the patient, using the Tasso+ device and blood collected in the office using a Vacutainer (SST, Red Top tube) using venipuncture for ALT, AST and total bilirubin, quantified using a Roche Cobas 8000/c702 or an equivalent analyzer.

SECONDARY OUTCOMES:
Venous and Tasso+ blood sample comparison for additional analytes | through study completion, an average of 1 Year and 6 Months
  Correlation of additional analytes including Total Protein, Albumin, Glucose, Sodium, Potassium, Chloride, Magnesium, Calcium, Phosphorus, Enzymatic Creatinine and alkaline Phosphatase (ALP) in blood collected with the Tasso+ device and by venipuncture in a Vacutainer (SST, Red Top tube) analyzed using a Roche Cobas 8000/c702 or an equivalent analyzer or an equivalent analyzer.
To collect patient experience with the Tasso blood collection | through study completion, an average of 1 Year and 6 Months
  To collect patient experience with the Tasso blood collection utilizing a brief survey aimed at understanding patient experience and preferences on the use and adoption of Tasso+ to collect a blood sample independently (with the help of a caregiver if needed), outside of the clinic.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - EvergreenHealth Research, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wickremsinhe E, Fantana A, Berthier E, Quist BA, Lopez de Castilla D, Fix C, Chan K, Shi J, Walker MG, Kherani JF, Knoderer H, Regev A, Harding JJ. Standard Venipuncture vs a Capillary Blood Collection Device for the Prospective Determination of Abnormal Liver Chemistry. J Appl Lab Med. 2023 May 4;8(3):535-550. doi: 10.1093/jalm/jfac127. PMID 36533519